CLINICAL TRIAL: NCT04341142
Title: Assessment of Serological Techniques for Screening Patients Regarding COVID-19-COVID-SER
Acronym: COVID-SER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL20_0329
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: CoV2 Positive Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serological tests will be applied on patients blood sampling (Experimental): Serological tests will be applied on patients blood sampling
  Interventions: Diagnostic Test: Serological tests will be applied on patients blood sampling

INTERVENTIONS:
Diagnostic Test: Serological tests will be applied on patients blood sampling — Application of tests on patients' serum

SUMMARY:
Covid-SER is a prospective multi-center study for the evaluation of diagnostic performance of available serological tests

ELIGIBILITY:
Inclusion Criteria:

* Seropositive caregivers screened for anti-SARS CoV2 antibodies during their consultation at the occupational medicine of HCL.
* Age: ≥ 18 years old
* Persons having given their written consent and accepting a follow-up every 6 months for 24 months, followed by a final visit at 36 months.
* Persons affiliated to a social security scheme or beneficiary of such a scheme.

Exclusion Criteria:

* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2020-04-10 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
The positivity (Yes/No) of the serological test. | Day 0
  The sensitivity and specificity of serological tests (positive or negative) compared to molecular detection of the virus by PCR
The positivity (Yes/No) of the serological test. | Day 3
  The sensitivity and specificity of serological tests (positive or negative) compared to molecular detection of the virus by PCR
The positivity (Yes/No) of the serological test. | Day 7
  The sensitivity and specificity of serological tests (positive or negative) compared to molecular detection of the virus by PCR
The positivity (Yes/No) of the serological test. | Day 14
  The sensitivity and specificity of serological tests (positive or negative) compared to molecular detection of the virus by PCR
The positivity (Yes/No) of the serological test. | Day 21
  The sensitivity and specificity of serological tests (positive or negative) compared to molecular detection of the virus by PCR
The positivity (Yes/No) of the serological test. | Day 28
  The sensitivity and specificity of serological tests (positive or negative) compared to molecular detection of the virus by PCR
The positivity (Yes/No) of the serological test. | Day 35
  The sensitivity and specificity of serological tests (positive or negative) compared to molecular detection of the virus by PCR
The positivity (Yes/No) of the serological test. | Day 42
  The sensitivity and specificity of serological tests (positive or negative) compared to molecular detection of the virus by PCR

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lyon Sud,Sainte Eugénie bat 4M,5, Chemin du Grand Revoyet, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bal A, Trabaud MA, Fassier JB, Rabilloud M, Saker K, Langlois-Jacques C, Guibert N, Paul A, Alfaiate D, Massardier-Pilonchery A, Pitiot V, Morfin-Sherpa F, Lina B, Pozzetto B, Trouillet-Assant S; COVID SER Study Group. Six-month antibody response to SARS-CoV-2 in healthcare workers assessed by virus neutralization and commercial assays. Clin Microbiol Infect. 2021 Jun;27(6):933-935. doi: 10.1016/j.cmi.2021.01.003. Epub 2021 Jan 13. No abstract available. PMID 33450388
- [Result] Bal A, Brengel-Pesce K, Gaymard A, Queromes G, Guibert N, Frobert E, Bouscambert M, Trabaud MA, Allantaz-Frager F, Oriol G, Cheynet V, d'Aubarede C, Massardier-Pilonchery A, Buisson M, Lupo J, Pozzetto B, Poignard P, Lina B, Fassier JB, Morfin F, Trouillet-Assant S; COVID-SER Study group. Clinical and laboratory characteristics of symptomatic healthcare workers with suspected COVID-19: a prospective cohort study. Sci Rep. 2021 Jul 22;11(1):14977. doi: 10.1038/s41598-021-93828-y. PMID 34294751
- [Result] Pozzetto B, Legros V, Djebali S, Barateau V, Guibert N, Villard M, Peyrot L, Allatif O, Fassier JB, Massardier-Pilonchery A, Brengel-Pesce K, Yaugel-Novoa M, Denolly S, Boson B, Bourlet T, Bal A, Valette M, Andrieu T, Lina B; Covid-Ser study group; Cosset FL, Paul S, Defrance T, Marvel J, Walzer T, Trouillet-Assant S. Immunogenicity and efficacy of heterologous ChAdOx1-BNT162b2 vaccination. Nature. 2021 Dec;600(7890):701-706. doi: 10.1038/s41586-021-04120-y. Epub 2021 Oct 21. PMID 34673755
- [Result] Trouillet-Assant S, Albert Vega C, Bal A, Nazare JA, Fascia P, Paul A, Massardier-Pilonchery A, D Aubarede C, Guibert N, Pitiot V, Lahousse M, Boibieux A, Makhloufi D, Simon C, Rabilloud M, Trabaud MA, Gueyffier F, Fassier JB; COVID-SER study group. Assessment of serological techniques for screening patients for COVID-19 (COVID-SER): a prospective, multicentric study. BMJ Open. 2020 Nov 24;10(11):e041268. doi: 10.1136/bmjopen-2020-041268. PMID 33234651
- [Result] de Boer J, Saade U, Granjon E, Trouillet-Assant S, Saade C, Pottel H, Zrein M; Covid ser study group. A novel assessment method for COVID-19 humoral immunity duration using serial measurements in naturally infected and vaccinated subjects. PLoS One. 2022 Sep 29;17(9):e0274553. doi: 10.1371/journal.pone.0274553. eCollection 2022. PMID 36173972
- [Result] Bal A, Pozzetto B, Trabaud MA, Escuret V, Rabilloud M, Langlois-Jacques C, Paul A, Guibert N, D'Aubarede-Frieh C, Massardier-Pilonchery A, Fabien N, Goncalves D, Boibieux A, Morfin-Sherpa F, Pitiot V, Gueyffier F, Lina B, Fassier JB, Trouillet-Assant S; COVID SER Study Group. Evaluation of High-Throughput SARS-CoV-2 Serological Assays in a Longitudinal Cohort of Patients with Mild COVID-19: Clinical Sensitivity, Specificity, and Association with Virus Neutralization Test. Clin Chem. 2021 Apr 29;67(5):742-752. doi: 10.1093/clinchem/hvaa336. PMID 33399823